CLINICAL TRIAL: NCT04724733
Title: Promoting Risk Reduction Among Young Adults With Asthma During Wildfire Smoke Events (TRAK)
Acronym: TRAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Julie Postma, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18035; 1R21NR019071-01 (NIH)
Record Dates: First submitted 2020-06-19; First posted 2021-01-26 (Actual); Results first posted 2022-08-02 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Asthma
Keywords: Young adult; quality of life; wildfires; risk reduction behavior; smartphone
MeSH Terms: conditions — Asthma; Pemphigus and fogo selvagem; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized with equal probability to 1 of 3 study groups in blocks of 2, 4 and 5. Random assignment of the participants will be determined using a randomization software. Random group assignment and a corresponding unique study identification (ID) number will be placed in sealed envelopes that are numbered sequentially. After the consent is signed, research personnel will open the envelope to reveal the participant's group assignment. Research personnel will record the participant's name, study ID and group assignment in a password-protected spreadsheet stored on a secure server at WSU. As part of (virtual) study visit 1, intervention participants will download the app to their smartphones. A set-up macro will ask the participant to enter their study ID which can be associated with all data captured by the app.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The control group will receive incentives for study participation but will not be introduced to the Smoke Sense app.
- Smoke Sense (Experimental)
  Interventions: Behavioral: Smoke Sense
- Smoke Sense Plus (Active Comparator)
  Interventions: Behavioral: Smoke Sense Plus

INTERVENTIONS:
Behavioral: Smoke Sense — Smoke Sense is a smartphone application (app). Smoke Sense participants will be asked to establish a profile which includes demographics, baseline health information and current beliefs about smoke and air pollution. In the Symptoms & Smoke Observations tab, participants are asked to report their weekly observations of smoke, health symptoms, and exposure reduction behaviors. In the Fire & Smoke Near Me tab, participants review the most recent AQ data measured at an AQ monitoring sites. Participants are asked to complete the AQ 101 module which test knowledge of AQ facts and provides correct answers. Badges are awarded for accomplishments within the app to promote certain desired behaviors: completing a user profile, launching the app weekly to check local AQ, reporting smoke and symptom observations, expanding AQ knowledge with AQ lessons, and exploring the map. Finally, participants can engage with other users by viewing cumulative statistics of symptoms and smoke observations.
  Arms: Smoke Sense
Behavioral: Smoke Sense Plus — Participants randomized to the Smoke Sense Plus intervention will be asked to do everything that the Smoke Sense intervention group does on a weekly basis, as well as: 1) Receive weekly push notifications that remind them to, for example, review their asthma action plan, refill any expired medications, take their daily controller medication, identify a clean air space in their home and community, 2) Monitor their lung function weekly via mobile spirometry, and 3) Subscribe to a social network to share strategies to minimize exposure.
  Arms: Smoke Sense Plus

SUMMARY:
This research will contribute to fundamental knowledge about how young adults with asthma perceive their personal health risks to wildfire smoke, minimize their risk, and improve their health. The investigators will compare young adults who use 'Smoke Sense,' an EPA-developed smart phone application (app), with young adults who use the app plus engage in preventive activities, with young adults who do not use the app. Study aims are to:

1. Establish the feasibility (recruitment, enrollment, retention rates), acceptability (intervention engagement, fidelity, usability, attitude) and barriers and facilitators of adopting the technology of the Smoke Sense interventions and use of portable devices in young adults with asthma;
2. Explore the preliminary impact of the Smoke Sense interventions on lung function and asthma control. These primary outcomes will be assessed using objective measures (spirometry) and validated, self-report tools.

   Secondary outcomes will be anxiety, exposure reduction behaviors (e.g. stayed indoors, wore a mask), and symptom mitigating behaviors (use of medication, unscheduled health care appointments), measured via self-report and a Global Positioning System device. Outcome by group will be summarized. Preliminary evidence of treatment effect and its variance will be examined for a future clinical trial;
3. Explore potential mediators (medication adherence, self-management skills, stress) and moderators (asthma severity/control) of the interventions to asthma outcomes. The long-term goal is to minimize asthma exacerbations from exposure to wildfire smoke.

The long-term goal of the study is to minimize asthma exacerbations from exposure to wildfire smoke.

DETAILED DESCRIPTION:
Exposure to unprecedented levels of wildfire smoke is increasing cardiopulmonary mortality and is especially catastrophic in people with asthma. Little evidence exists on the effectiveness of air quality (AQ) alerts on objective measures of risk reduction behavior and health outcomes. Evidence shows that young adults are less likely to adhere to AQ alerts than older adults, yet young adulthood is a time when habits are formed in chronic illness management. The Environmental Protection Agency's (EPA) Smoke Sense smart phone application (app) is an innovative risk reduction intervention based on the health belief model and theory of planned behavior. The app invites users to record their smoke observations and health symptoms, play educational trivia games, earn badges, and explore what other users are reporting. Smoke Sense connects AQ exposure data with users' symptoms, thus framing risk reduction messages as personally relevant. Although Smoke Sense has almost 25,000 users, its impact on health outcomes has not been tested. Preliminary data suggests that users' engagement in health protective behaviors was driven in response to symptoms rather than as preventive courses of action. In a high-risk asthma population, prevention is paramount. Smoke Sense Plus is an intervention that builds on the Smoke Sense app, with value-added activities, such as notifying participants to review their asthma action plan, monitoring lung function weekly via mobile spirometry and subscribing to a social network to share strategies to minimize exposure. The purpose of this study is to assess the feasibility of the Smoke Sense interventions among young adults with asthma and pilot test the interventions compared to a control group. Sixty young adults aged 18-26 with asthma will be recruited through local universities. They will be randomized to 1 of 3 groups for a 2-month study period during wildfire season. Study aims are to:

1. Establish the feasibility (recruitment, enrollment, retention rates), acceptability (intervention engagement, fidelity, usability, attitude) and barriers and facilitators of adopting the technology of the Smoke Sense interventions and use of portable devices in young adults with asthma;51
2. Explore the preliminary impact of the Smoke Sense interventions on lung function,20 and asthma control, These primary outcomes will be assessed using objective measures (spirometry) and validated, self-report tools. Secondary outcomes will be anxiety,23 exposure reduction behaviors (e.g. stayed indoors, wore a mask),24 and symptom mitigating behaviors (use of medication, unscheduled health care appointments), measured via self-report and a Global Positioning System device. Outcome by group will be summarized. Preliminary evidence of treatment effect and its variance will be examined for a future clinical trial;
3. Explore potential mediators (medication adherence, self-management skills, stress) and moderators (asthma severity/control) of the interventions to asthma outcomes. The long-term goal is to minimize asthma exacerbations from exposure to wildfire smoke.

The long-term goal of the study is to minimize asthma exacerbations from exposure to wildfire smoke.

ELIGIBILITY:
Inclusion Criteria:

* 18-26 years old
* Diagnosed with asthma by a health care provider
* Own a smart phone (Android or iOS platforms)
* Speak and read English

Exclusion Criteria:

* Already use the Smoke Sense app
* Had surgery within 3 weeks of the study start date
* Have a cardio-vascular condition
* Smoke
* Have or have had COVID 19 (that you're aware of)

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Postma, PhD, Principal Investigator — Washington State University College of Nursing
Locations (1):
- Washington State University College of Nursing, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Postma JM, Odom-Maryon T, Rappold AG, Haverkamp H, Amiri S, Bindler R, Whicker J, Walden V. Promoting risk reduction among young adults with asthma during wildfire smoke: A feasibility study. Public Health Nurs. 2022 Mar;39(2):405-414. doi: 10.1111/phn.12986. Epub 2021 Oct 11. PMID 34636066

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Smoke Sense | Smoke Sense Plus
Started | 22 | 22 | 23
4 Weeks | 22 | 21 | 23
Completed | 21 | 21 | 22
Not Completed | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Smoke Sense | Smoke Sense Plus | Total
Number analyzed (Participants) | 22 | 22 | 23 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 23 | 67
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (2.5) | 21.8 (2.81) | 21.9 (2.05) | 21.9 (2.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 17 | 51
  Male | 4 | 6 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 17 | 17 | 18 | 52
  More than one race | 3 | 3 | 2 | 8
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 23 | 67
asthma control test [Mean (Standard Deviation); unit: units on a scale] | 20.3 (3.4) | 20.7 (1.8) | 20.3 (2.2) | 20.4 (2.5)
mean percent predicted FEV1 [Mean (Standard Deviation); unit: percent] | 89.8 (20.1) | 96.2 (14.1) | 93.4 (18.6) | 93.1 (17.8)

OUTCOME MEASURES:

1. Primary Outcome: Lung Function, Specifically % Predicted Mean FEV1
Description: Lung function indicates future risk of adverse outcomes and is regularly monitored in people with asthma. Spirometry is used to objectively measure and monitor airway obstruction by blowing into a machine and measuring forced expiratory volume (FEV1), forced vital capacity (FVC), and their ratio (FEV1/FVC). A low FEV1, <60% predicted, is a potentially modifiable independent risk factor for severe asthma exacerbations. Portable spirometers, that are used by patients independently and connect to smartphones, have been validated against conventional spirometry performed by specialists in clinical settings.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of predicted
Arm/Group | Control | Smoke Sense | Smoke Sense Plus
Number analyzed (Participants) | 13 | 7 | 17
percentage of predicted | 92.9 (16) | 95.6 (17.2) | 88.6 (17.2)
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p > 0.05, t-test, 1 sided
Statistical Analysis 2: Comparison: Smoke Sense; Test type: Superiority; p > 0.05, t-test, 1 sided
Statistical Analysis 3: Comparison: Smoke Sense Plus; Test type: Superiority; p = 0.0172, t-test, 1 sided

2. Primary Outcome: Asthma Control Test
Description: The Asthma Control Test (ACT) measures the frequency of shortness of breath and general asthma symptoms, use of rescue medications, effect of asthma on daily functioning, and an overall self-assessment of asthma control via self-report. It has 5 items, is based on self report of symptoms and daily functioning and has a response scale that ranges from 5 (poor control) to 25 (complete control). ACT score >19 indicates well-controlled (versus 19 or < poorly controlled) asthma. The Minimally Important Difference (MID) is 3 points between two groups or for changes over time.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Smoke Sense | Smoke Sense Plus
Number analyzed (Participants) | 13 | 7 | 17
score on a scale | 22.4 (1.9) | 21 (4) | 21.5 (2.3)
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p = .0320, t-test, 1 sided
Statistical Analysis 2: Comparison: Smoke Sense; Test type: Superiority; p > 0.05, t-test, 1 sided
Statistical Analysis 3: Comparison: Smoke Sense Plus; Test type: Superiority; p = 0.0008, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: From consent throughout the 8 week study period.
Arm/Group | Control | Smoke Sense | Smoke Sense Plus
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/23

LIMITATIONS AND CAVEATS:
37 participants recorded both ACT and FEV1 measures that were within the study visit window (3 days from scheduled) and within 1 day of each other at both baseline and week 8. This limited our ability to assess changes in clinical outcomes and will be addressed in future work.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT04724733/Prot_SAP_ICF_000.pdf